CLINICAL TRIAL: NCT04733040
Title: A Phase IIa, Open-Label, 2-Arm Multicenter Clinical Trial to Evaluate the Efficacy, Safety and PK/PD of the Human Anti-CD38 Antibody MOR202 in Anti-PLA2R Antibody Positive Membranous Nephropathy (NewPLACE)
Brief Title: Efficacy, Safety and PK/PD of MOR202 in Anti-PLA2R+ Membranous Nephropathy (aMN) (NewPLACE)
Acronym: NewPLACE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HI-Bio, A Biogen Company (Industry)
Responsible Party: Sponsor
Organization: Biogen (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOR202C205
Record Dates: First submitted 2021-01-18; First posted 2021-02-01 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Glomerulonephritis; Membranous Nephropathy; antiPLA2R Positive
MeSH Terms: conditions — Glomerulonephritis; Glomerulonephritis, Membranous | interventions — felzartamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- MOR202 5 Doses (Experimental): 5 doses administered on Day 1, 8, 15, 29, and 57
  Interventions: Drug: MOR202
- MOR202 2 Doses (Experimental): 2 doses administered on Day 1 and 15
  Interventions: Drug: MOR202

INTERVENTIONS:
Drug: MOR202 — MOR202 will be administered as an intravenous infusion
  Other Names: Felzartamab

SUMMARY:
This 2-arm, multi-center, open-label, parallel-group phase II trial will assess the efficacy, safety and pharmacokinetics/pharmacodynamics of the human antibody MOR202 in subjects with anti-PLA2R antibody-positive membranous nephropathy indicated for immunosuppressive therapy

DETAILED DESCRIPTION:
After treatment, subjects will enter a repeat treatment period (3 months) if necessary; and a final follow-up period of 15 to 18 months.

Study Sponsor, originally HI-Bio, Inc., is now HI-Bio, A Biogen Company.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 18 to ≤ 80 years (at date of signing the informed consent form [ICF]).
* Urine protein to creatinine ratio (UPCR) of ≥ 3.0 g/g or proteinuria ≥ 3.5 g/24 h
* Estimated glomerular filtration rate (eGFR) ≥ 50 ml/min/1.73 m² (eGFR >30 and < 50 ml/min/1.73 m² can be included provided an interstitial fibrosis and tubular atrophy (IFTA) score of < 25% in a kidney biopsy)
* Not in spontaneous remission despite proper treatment with angiotensin-converting enzyme inhibitors (ACEI), angiotensin receptor blockers (ARBs) (sufficient dose and treatment duration) as per clinical practice and scientific guidelines. If the subject is intolerant to ACEI and ARBs, the reason must be documented and approval for enrollment be obtained from the Medical Monitor.
* Systolic blood pressure (BP) ≤150 mmHg and diastolic BP ≤100 mmHg after 5 minutes of rest.
* Serum anti-PLA2R antibodies ≥ 50.0 RU/mL determined by Euroimmun ELISA.
* Female subjects: A female is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  1. Not a female of childbearing potential (FCBP)
  2. A FCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 3 months after the last dose of MOR202

Key Exclusion Criteria:

* Hemoglobin < 80 g/L.
* Thrombocytopenia: Platelets < 100.0 x 10^9/L.
* Neutropenia: Neutrophils < 1.5 x 10^9/L.
* Leukopenia: Leukocytes < 3.0 x 10^9/L.
* Hypogammaglobulinemia: Serum immunoglobulins ≤ 4.0 g/L.

Subjects may receive supportive therapies to meet the above criteria

* B-cells < 5 x 10^6/L
* Diabetes mellitus type 2: Subjects with type 2 diabetes mellitus may only enter the clinical trial if a kidney biopsy performed within 6 months prior to screening shows MN without evidence of diabetic nephropathy and diabetes is controlled, as shown by:

  1. Glycated hemoglobin (HbA1c) <8.0 % or 64 mmol/mol.
  2. No diabetic retinopathy known.
  3. No peripheral neuropathy known.
* Total bilirubin, aspartate aminotransferase or alanine aminotransferase >1.5 x ULN, alkaline phosphatase >3.0 x ULN.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
efficacy: percent change of anti-PLA2R antibody levels | 3 months compared to baseline
  efficacy of 2 different dosing regimens of MOR202 in subjects with anti-PLA2R antibody positive MN

SECONDARY OUTCOMES:
efficacy: immunological complete response (ICR) rate | ICR rate at 3 months, 6 months, 12 months and 24 months
  efficacy of 2 different dosing regimens of MOR202
efficacy: overall proteinuria response (OPR) rate | OPR rate at 6 months, 12 months and 24 months.
  efficacy of 2 different dosing regimens of MOR202
safety: determined by the frequency, incidence and severity of TEAEs | through treatment completion, an average of 3 months per treatment period
  frequency, incidence and severity of treatment-emergent adverse events
PK profile | through study completion, an average of 1 year
  MOR202 serum concentrations after multiple i.v. administrations
immunogenicity | through study completion, an average of 1 year
  number of subjects developing anti-MOR202 antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — HI-Bio, A Biogen Company
Locations (25):
- Georgia (2):
  - Managadze National Center of Urology, Tbilisi
  - Tbilisi State Medical University and Ingorokva High Medical Technology University Clinic, Tbilisi
- Germany (5):
  - University Hospital Aachen, Aachen
  - Charite, Berlin
  - DaVita Clinical Research, Düsseldorf
  - Uniklinikum, Essen
  - Hospital of Johannes Gutenberg University, Mainz
- Greece (4):
  - General Hospital of Athens, Athens
  - General Hospital of Heraklion Venizeleio-Papaneio, Heraklion
  - University General Hospital of Patras, Pátrai
  - General Hospital of Thessaloniki, Thessaloniki
- Russia (2):
  - Botkin Hospital Moscow, Moscow
  - First Pavlov State Medical University of St. Petersburg, Saint Petersburg
- South Korea (5):
  - Hallym University Sacred Heart Hospital, Chuncheon
  - JeJu National University Hospital, Jeju City
  - Konkuk University Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Seoul National University Bundang Hospital, Seoul
- Taiwan (5):
  - Chang Gung Memorial Hospital, Kaohsiung City
  - Shuang Ho Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- United Kingdom (2):
  - Kings College, London
  - Nottingham Renal and Transplant Unit, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- [Derived] Ahmad SB, Jefferson JA. Targeting B Cells and Plasma Cells in Glomerular Disease. J Am Soc Nephrol. 2025 Jun 4;36(9):1844-1857. doi: 10.1681/ASN.0000000772. PMID 40465397